CLINICAL TRIAL: NCT04256876
Title: A Randomized-controlled Trial Comparing Transcutaneous Tibial Nerve Stimulation (TTNS) Versus Sham Therapy on Short Term Continence Outcomes in Children With the Idiopathic Overactive Bladder Syndrome: the TaPaS Trial Part I
Brief Title: TTNS Versus Sham Therapy for Children With iOAB (TaPaS Part I)
Acronym: TaPaS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the corona pandemic, live patient contact was no longer possible. As a result, the study had to be stopped early.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC/2018/1267
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective randomized-controlled superiority trial:
  TTNS(Active treatment) vs. Sham TTNS (placebo)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded for the given treatment ( Active TTNS vs. Sham TTNS) by the care provider ( Physiotherapist).
  The outcomes assessor (the pediatric urologist) isn't aware of the treatment neither.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active TTNS (Active Comparator): Children treated by transcutaneous tibial nerve stimulation. TENS device connected to adhesive electrodes. Stimulation settings: 200 µS, 20 Hz, 1-20 V ( depending of sensory response) Home-therapy: Daily stimulation during 60 minutes.
  Interventions: Device: TTNS
- TTNS sham intervention (Sham Comparator): Children treated by TTNS with same positioning as the active TTNS treatment. Stimulation settings: 200 µS, 20 Hz, 0-1 V. Patients and parents will be told that electric currence is given, but that no sensation will be feld.
  Home therapy: Daily stimulation during 60 minutes.
  Interventions: Device: TTNS Sham

INTERVENTIONS:
Device: TTNS — See section 'arms' Stimulation settings: 200 µS, 20 Hz, 1-20 V ( depending of sensory response) Home-therapy: Daily stimulation during 60 minutes.
  Other Names: Transcutaneous tibial nerve stimulation
  Arms: Active TTNS
Device: TTNS Sham — See section 'arms'
  Other Names: Sham therapy
  Arms: TTNS sham intervention

SUMMARY:
Part I of the TaPaS trial forms part of a twofold clinical RCT:

Part 1) A prospective RCT comparing the efficacy of transcutaneous tibial nerve stimulation (TTNS) with TTNS sham therapy for children with idiopathic overactive bladder on clinical and patient reported outcomes (PROMS).

Part 2) A prospective RCT comparing TTNS versus Percutaneous tibial nerve stimulation (PTNS) on clinical outcomes and PROMS.

DETAILED DESCRIPTION:
Non invasive neuromodulation therapy for children with the overactive bladder syndrome is a highly under investigated topic in medical literature.

Only 2 studies ( Patidar et al. and Boudaouid et al.) investigated the use of tibial nerve stimulation with adhesive electrodes.

1) In the first trial the superiority of TTNS vs.Sham therapy for the therapeutic management of children with OAB naive to any pharmacological treatment will be examined.

Clinical outcomes will be assessed by the use of daytime and nighttime bladder diaries.

Assessment of outcomes at baseline, after 6 weeks and 12 weeks of treatment, and investigation of mean time to partial or complete relapse following 6 weeks observation.

After a wash-out period of 6 weeks, patients from the part I Sham group will be able to be included for TaPaS part II.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5 and 12 years old, clinically diagnosed with the idiopathic overactive bladder syndrome with urinary incontinence (daytime and/or nighttime)
* Untreated, except from urotherapy.

Exclusion Criteria:

* Enuresis nocturna due to nocturnal polyuria
* Dysfunctional voiding
* Neurogenic bladder
* Psychiatric disorders, behavioural disturbances or mental disabilities
* Treated before with pharmacotherapy or invasive therapies for OAB
* Children with parents unable to record reliably micturition diaries.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Mean voided volume per void | 12 weeks
  Difference in mean voided volume per void in percentage

SECONDARY OUTCOMES:
Maximum voided volume (ml) | 12 weeks
  Maximal voided volume per void ( ml) .
Number of urgency incontinence episodes / 24 h. | 12 weeks
  Reduction in number of incontinence episodes per 24 hour
Daytime voiding frequency | 12 weeks
  Mean voiding frequency per day
Satisfaction on urinary symptoms reported by parents | 12 weeks
  Subjective satisfaction reported by the parents - on a 7 point likert scale- "How satisfied of dissatisfied would you be if the bladder symptoms of your child would persist like this?
Time to recurrence | At 12 weeks of treatment + at 6 weeks of observational period without treatment.
  Time to complete or partial relapse to baseline symptoms after 12 weeks of treatment during the observational period of 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Spinoit, Professor, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boudaoud N, Binet A, Line A, Chaouadi D, Jolly C, Fiquet CF, Ripert T, Merol ML. Management of refractory overactive bladder in children by transcutaneous posterior tibial nerve stimulation: A controlled study. J Pediatr Urol. 2015 Jun;11(3):138.e1-10. doi: 10.1016/j.jpurol.2014.09.013. Epub 2015 Mar 31. PMID 25979217
- [Result] Patidar N, Mittal V, Kumar M, Sureka SK, Arora S, Ansari MS. Transcutaneous posterior tibial nerve stimulation in pediatric overactive bladder: A preliminary report. J Pediatr Urol. 2015 Dec;11(6):351.e1-6. doi: 10.1016/j.jpurol.2015.04.040. Epub 2015 Jul 29. PMID 26279104
- [Derived] Ghijselings L, Renson C, Van de Walle J, Everaert K, Spinoit AF. Clinical efficacy of transcutaneous tibial nerve stimulation (TTNS) versus sham therapy (part I) and TTNS versus percutaneous tibial nerve stimulation (PTNS) (part II) on the short term in children with the idiopathic overactive bladder syndrome: protocol for part I of the twofold double-blinded randomized controlled TaPaS trial. Trials. 2021 Apr 2;22(1):247. doi: 10.1186/s13063-021-05117-8. PMID 33810804